CLINICAL TRIAL: NCT05057013
Title: A Cancer Research UK Phase I/IIa Open Label, Dose Escalation and Expansion Trial of HMBD-001 (an Anti-HER3 Monoclonal Antibody) Given Intravenously as a Single Agent and in Combination in Patients With Advanced HER3 Positive Solid Tumours
Brief Title: A Phase I/IIa Trial of HMBD-001 in Advanced HER3 Positive Solid Tumours
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cancer Research UK (Other)
Collaborators: Hummingbird Bioscience (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRUKD/22/002; 2020-005891-36 (EudraCT Number)
Record Dates: First submitted 2021-09-10; First posted 2021-09-27 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Bladder Cancer; Triple Negative Breast Cancer; Castration-resistant Prostate Cancer; Cervical Cancer; RAS Wild Type Colorectal Cancer; Endometrial Cancer; Gastric Cancer; Hepatocellular Carcinoma (HCC); Melanoma; Non-small Cell Lung Cancer (NSCLC); Oesophageal Cancer; Ovarian Cancer; Pancreatic Cancer; Squamous Cell Cancer of the Head and Neck
Keywords: Antibodies, monoclonal; HER3; Receptor, ErbB-3; NRG1; NRG1 gene fusion; Neuregulin 1; Androgen receptor antagonists; Prostatic neoplasms, castration-resistant
MeSH Terms: conditions — Urinary Bladder Neoplasms; Triple Negative Breast Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms; Stomach Neoplasms; Carcinoma, Hepatocellular; Melanoma; Carcinoma, Non-Small-Cell Lung; Esophageal Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms; Lethal Congenital Contracture Syndrome 2; Fibromatosis, Gingival, 2; Prostatic Neoplasms, Castration-Resistant | interventions — enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HMBD-001 (Part A) (Experimental)
  Interventions: Drug: HMBD-001
- HMBD-001 and enzalutamide (Part B Arm 1) (Experimental)
  Interventions: Drug: HMBD-001 and enzalutamide

INTERVENTIONS:
Drug: HMBD-001 — Participants with advanced solid tumours will receive their assigned dose level of HMBD-001 diluted in 0.9% sodium chloride, administered once a week as a 120-minute intravenous (IV) infusion. Cycles are 28 days with no break in between; administration may continue for up to 6 cycles but may continue for longer if the participant is deemed to be benefitting.
  Arms: HMBD-001 (Part A)
Drug: HMBD-001 and enzalutamide — Participants with metastatic castration resistant prostate cancer (mCRPC) confirmed as HER3 positive with no PTEN loss or with a NRG1 fusion rearrangement will receive the HMBD-001 recommended Phase 2 dose (RP2D) as determined in Part A, diluted in 0.9% sodium chloride and administered once a week as a 120-minute IV infusion, in combination with enzalutamide administered at a fixed dose of 160 mg once daily, in 28-day cycles with no break between cycles. Immediately before commencing combination therapy, participants may receive one 28-day cycle of enzalutamide monotherapy to confirm that their disease does not respond to enzalutamide alone. HMBD-001 may be administered for up to 6 cycles; enzalutamide may be continued until disease progression or unacceptable toxicity.
  Arms: HMBD-001 and enzalutamide (Part B Arm 1)

SUMMARY:
This clinical trial is evaluating a drug called HMBD-001 (an anti-HER3 monoclonal antibody) in participants with advanced HER3 positive solid tumours. The main aims are to find out the best dose of HMBD-001 that can be given to participants alone and in combination with other anti-cancer agents, more about the potential side effects of HMBD-001 and how they can be treated, and what happens to HMBD-001 inside the body and how it affects cancer cells.

DETAILED DESCRIPTION:
HMBD-001 is a type of drug called a monoclonal antibody. It works by targeting a protein called HER3, which is found in high numbers in some types of cancers including those that contain fusions in a gene called NRG1. By attaching itself to this protein, it may then work to kill the cancer cells or to stop them growing.

This is a first-in-human clinical trial that has two parts:

Part A is a 'dose escalation' phase where small groups of participants will receive increasing doses of HMBD-001 on its own (as a single agent) to find the safest dose that best targets cancer cells.

Part B is a 'dose expansion' phase where larger groups of participants with specific cancer types that are known to have high levels of the protein HER3 or that have a confirmed NRG1 gene fusion will receive the highest doses of HMBD-001 considered to be safe as monotherapy from Part A in combination with other anti-cancer drugs that are already licensed for use.

In Part B Arm 1, participants will receive HMBD-001 in combination with enzalutamide. Enzalutamide is a drug used to treat prostate cancer. Prostate cancer is known to be sensitive to androgens (hormones associated with male characteristics), and enzalutamide blocks the action of androgens by limiting the binding of androgens to androgen receptors. This slows the growth of prostate cancer cells and may kill them.

The main aims of the clinical trial are to find out:

* The best dose of HMBD-001 alone and in combination with other anti-cancer drugs that should be given to participants.
* More about the potential side effects of HMBD-001 when given alone and in combination with other anti-cancer agents, and how they can be managed.
* What happens to HMBD-001 inside the body and how it affects cancer cells.
* The potential anti-tumour activity of HMBD-001 as a single agent and in combination with other anti-cancer agents in specific tumour types of HER3-expressing tumours or tumours with NRG1 gene fusions.

ELIGIBILITY:
Inclusion criteria:

1. Written (signed and dated) informed consent and be capable of co-operating with HMBD-001 administration and follow-up.
2. Part A: Monotherapy Dose Escalation

   Histologically confirmed advanced or metastatic solid tumours resistant or refractory to conventional treatment, or for which no conventional therapy exists or is not considered appropriate by the Investigator or is declined by the participant.

   Participants with tumour types known to overexpress HER3 including:
   * Bladder cancer
   * Triple negative breast cancer
   * Castration resistant prostate cancer
   * Cervical cancer
   * RAS wild type colorectal cancer
   * Endometrial cancer
   * Gastric cancer
   * Hepatocellular carcinoma (HCC)
   * Melanoma
   * Non-small cell lung cancer (NSCLC)
   * Oesophageal cancer
   * Ovarian cancer
   * Pancreatic cancer
   * Squamous cell cancers of the head and neck

   Participants with a confirmed existing NRG1 fusion rearrangement or HER amplification will also be considered eligible.

   Part B Arm 1: HMBD-001 and Enzalutamide Combination
   * Histologically confirmed metastatic castration-resistant prostate adenocarcinoma without neuroendocrine differentiation or small-cell features.
   * Serum testosterone concentration ≤50 ng/dL sustained by medical or surgical castration.
   * Participants must have progressive disease prior to study enrolment.
   * PSA at screening ˃1 ng/mL.
   * Confirmed high HER3 expression.
   * Absence of PTEN loss.
   * Participants with confirmed existing NRG1 fusion rearrangement will also be considered eligible.
3. Life expectancy of at least 12 weeks.
4. Eastern Cooperative Oncology Group performance status of 0 or 1.
5. Haematological and biochemical indices within the protocol specified ranges.
6. Participants with advanced prostate cancer must have castrate levels of testosterone and have received a next generation hormonal agent (at least one of abiraterone, enzalutamide, apalutamide or darolutamide).
7. Part A: Aged 16 years or over at the time consent is given.
8. Part B Arm 1: Aged 18 years or over at the time consent is given.

Exclusion criteria

1. Radiotherapy (except for palliative reasons), chemotherapy, endocrine therapy (with the exception of life-long hormone suppression such as luteinising hormone-releasing hormone agents in prostate cancer), immunotherapy or investigational medicinal products during the previous 4 weeks before first dose of HMBD-001 or enzalutamide, as applicable.
2. Participants with ongoing toxic manifestations of previous treatments greater than NCI CTCAE Grade 1. Exceptions apply.
3. Participants with symptomatic brain or leptomeningeal metastases should be excluded. Exceptions apply.
4. Women of child-bearing potential (or are already pregnant or lactating). Exceptions apply.
5. Male participants with partners of child-bearing potential. Exceptions apply.
6. Major surgery from which the participant has not yet recovered.
7. At high medical risk because of non-malignant systemic disease including active uncontrolled infection.
8. Known to be serologically positive for hepatitis B, hepatitis C or human immunodeficiency virus infection. Participants with previous hepatitis C exposure but no current infection are eligible to participate.
9. Known or suspected hypersensitivity reaction to previous biological therapy that in the opinion of the Investigator is a contraindication for their participation in this study.
10. Concurrent congestive heart failure, prior history of ≥ Class II cardiac disease (New York Heart Association), clinically significant cardiac ischaemia or clinically significant cardiac arrhythmia. Participants with significant cardiovascular disease as defined in the protocol are excluded.
11. Active autoimmune disease. Exceptions apply.
12. Participants receiving doses of prednisolone ˃10 mg daily (or equipotent doses of other corticosteroids) within 7 days prior to the first dose of study drug are not eligible unless administered as pre-medication.
13. Participants having received a live vaccination within 4 weeks prior to first dose of HMBD-001.
14. Is a participant or plans to participate in another interventional clinical trial, whilst taking part in this Phase 1/2a trial of HMBD-001. Participation in an observational trial or interventional clinical trial which does not involve administration of an IMP and which would not place an unacceptable burden on the participant in the opinion of the Investigator and Medical Advisor would be acceptable.
15. Any other condition which in the Investigator's opinion would not make the participant a good candidate for the clinical trial.
16. Current or prior malignancy which could affect safety or efficacy assessment of the IMP or compliance with the protocol or interpretation of results. Participants with curatively-treated non-melanoma skin cancer, non-muscle-invasive bladder cancer, or carcinomas-in-situ are generally eligible.

    Part B Arm 1: HMBD-001 and Enzalutamide Combination:
17. Participants receiving warfarin or coumarin-like anti-coagulants.
18. History of seizures or other risk factors for the development of seizures e.g. prior history of stroke, brain injury, brain metastases, leptomeningeal disease.
19. Participants with hypersensitivity to enzalutamide or any of the excipients
20. Participants who have received prior enzalutamide or other next generation hormonal agent that has been stopped due to toxicities or intolerance or required a dose reduction during administration due to toxicity or intolerance.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2021-11-10 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Experienced Dose Limiting Toxicities (DLTs); Part A | From first dose onwards until completion of Cycle 1 (28 days)
  DLTs graded for severity using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0, measured by count of participants per arm.
Number of Participants Who Experienced DLTs; Part B Arm 1 | From first dose of combination therapy onwards until completion of Cycle 1 (28 days)
  DLTs graded for severity using the NCI CTCAE v5.0, measured by count of participants per arm.
Number of adverse events (AEs) by arm considered to be at least possibly related to HMBD-001 (Part A and Part B Arm 1) | From the date of written informed consent until the end of the safety follow-up period (maximum [max] 42 weeks per participant)
  Number of AEs related to HMBD-001 given as a single agent and in combination with enzlutamide, graded according to NCI CTCAE v5.0.
Number of Grade 3, 4 and 5 AEs by arm considered to be at least possibly related to HMBD-001 (Part A and Part B Arm 1) | From the date of written informed consent until the end of the safety follow-up period (max 42 weeks per participant)
  Number of Grade 3, 4 and 5 AEs related to HMBD-001 given as a single agent and in combination with enzalutamide, graded according to NCI CTCAE v5.0.
Overall response rate (ORR) within 6 cycles of HMBD-001 (Part B Arm 1) | From baseline radiological disease assessment until 28 days after last dose of HMBD-001 (max 36 weeks per participant)
  Proportion of participants who achieve a best response of complete response (CR) or partial response (PR), based on Response Evaluation Criteria in Solid Tumours (RECIST) v1.1 and/or Prostate Cancer Working Group 3 (PCWG3) Criteria as applicable, within 6 cycles of HMBD-001 in combination with enzalutamide.

SECONDARY OUTCOMES:
ORR within 6 cycles of HMBD-001 (Part A) | From baseline radiological disease assessment until 28 days after last dose of HMBD-001 (max 32 weeks per participant)
  Proportion of participants who achieve a best response of CR or PR, based on RECIST v1.1 and/or PCWG3 Criteria as applicable, within 6 cycles of HMBD-001 monotherapy.
Maximum observed serum concentration (Cmax) of HMBD-001 (Part A and Part B Arm 1) | Up to 31 timepoints from first dose until 28 days after the last dose of HMBD-001 (max 28 weeks per participant)
  Cmax of HMBD-001 in serum, analysed via enzyme linked immunosorbent assay (ELISA). Not all participants will be analysed at all timepoints.
Minimum observed serum concentration (Cmin) of HMBD-001 (Part A and Part B Arm 1) | Up to 31 timepoints from first dose until 28 days after the last dose of HMBD-001 (max 28 weeks per participant)
  Cmin of HMBD-001 in serum, analysed via ELISA. Not all participants will be analysed at all timepoints.
Area under the serum concentration-time curve (AUC) of HMBD-001 (Part A and Part B Arm 1) | Up to 31 timepoints from first dose until 28 days after the last dose of HMBD-001 (max 28 weeks per participant)
  AUC of HMBD-001, analysed via ELISA. Not all participants will be analysed at all timepoint
Terminal elimination half-life (t½) of HMBD-001 (Part A and Part B Arm 1) | Up to 31 timepoints from first dose until 28 days after the last dose of HMBD-001 (max 28 weeks per participant)
  t½ of HMBD-001 in serum, analysed via ELISA. Not all participants will be analysed at all timepoints.
Steady state volume of distribution of HMBD-001 in serum (Part A and Part B Arm 1) | Up to 31 timepoints from first dose until 28 days after the last dose of HMBD-001 (max 28 weeks per participant)
  Volume of distribution of HMBD-001 in serum at steady state, analysed via ELISA. Not all participants will be analysed at all timepoints.
Total body clearance of HMBD-001 (Part A and Part B Arm 1) | Up to 31 timepoints from first dose until 28 days after the last dose of HMBD-001 (max 28 weeks per participant)
  Total body clearance of HMBD-001 measured in serum, analysed via ELISA. Not all participants will be analysed at all timepoints.
ORR within 8 and 16 weeks of commencing HMBD-001 (Part A and Part B Arm 1) | From baseline radiological disease assessment up to 16 weeks post first HMBD-001 administration (max 24 weeks per participant)
  Proportion of participants achieving a best response of CR, or PR according to RECIST v1.1 and/or PCWG3 Criteria as applicable, within 8 and 16 weeks of commencing HMBD-001 as monotherapy and in combination with enzalutamide.
Disease control rate within 6 cycles of HMBD-001 (Part A and Part B Arm 1) | From baseline radiological disease assessment up to 28 days post last HMBD-001 administration (max 36 weeks per participant)
  Proportion of participants achieving a best response of CR, PR or stable disease (SD), based on RECIST v1.1 and/or PCWG3 Criteria as applicable, within 6 cycles of HMBD-001 as monotherapy and in combination with enzalutamide.
Duration of response (Part A and Part B Arm 1) | From the date of first recorded response until 24 months after the last enrolled participant's first dose of HMBD-001 (max 48 months per participant)
  The median duration in days from the first observation of a CR or PR, according to RECIST v1.1 and/or PCWG3 Criteria as applicable, until either progressive disease (PD) or death from any cause, in participants with a confirmed CR or PR.
Duration of clinical benefit (Part A and Part B Arm 1) | From the date of first recorded response until 24 months after the last enrolled participant's first dose of HMBD-001(max 48 months per participant)
  The median duration in days from the first administration of HMBD-001 until either PD or death from any cause, in participants who achieve a CR, PR, or SD for at least 24 weeks, according to RECIST v1.1 and/or PCWG3 Criteria as applicable.
Progression free survival (Part B Arm 1) | From first dose of HMBD-001 until 24 months after the last enrolled participant's first dose of HMBD-001 (max 48 months per participant)
  The median duration in days from first dose of HMBD-001 to death from any cause or PD according to RECIST v1.1 and/or PCWG3 Criteria as applicable.
Overall survival (Part B Arm 1) | From first dose of HMBD-001 until 24 months after the last enrolled participant's first dose of HMBD-001 (max 48 months per participant)
  The median time from first dose of HMBD-001 to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Johann de Bono, Prof, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (4):
- United Kingdom (4):
  - Royal Marsden NHS Foundation Trust, London
  - The Christie Hospital, Manchester
  - Freeman Hospital, Newcastle, Newcastle
  - Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No